CLINICAL TRIAL: NCT06976073
Title: Non-invasive Imaging for In-vivo Quantification of Skin Composition and Structure
Acronym: Spectrum1
Status: Recruiting | Type: Observational
Sponsor: HJN Sverige AB/Neko Health (Industry)
Responsible Party: Sponsor
Other Study IDs: TCI-P3-LMV_220623; CIV-22-07-039907 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2023-07-28; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Foot; Peripheral Arterial Disease; Skin Cancer; Cardiovascular Disease Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Foot; Peripheral Arterial Disease; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient_cohort: Adult patients mainly from a primary care cohort. All patients visiting the clinical sites, seeking care, or as separately invited, are offered to participate in this investigation. This includes sub-groups of patients with conditions such as diabetes mellitus, peripheral arterial disease and skin cancer. All participants undergo at least one examination with the investigational device (TCI P3).

SUMMARY:
The goal of this clinical investigation is to explore a non-invasive technology for measuring the microcirculatory structure, composition and function in patients from a primary care population.

The main aims are:

1. To evaluate the robustness of the technology for assessment of the molecular composition and structure of the skin tissue and microcirculatory function, on a prospective primary care population.
2. To evaluate the device and method on its capability to detect deficiencies in circulation, compared with existing reference systems with similar characteristics for patients with known cardiovascular disease risk and/or diabetes.

DETAILED DESCRIPTION:
The clinical investigation aims to evaluate the potential value of an investigational medical device (IMD) based on a technology called SFDI, Spatial Frequency Domain Imaging. This is a non-invasive contactless technology for in-vivo measurement of the structure and molecular composition of the skin and its embedded blood volume. The technology is a promising tool for diagnostic support of pathology to the microcirculation, like in peripheral arterial disease and diabetes, but also for general cardiovascular disease risk assessment.

The IMD can measure the concentration of deoxy- and oxyhemoglobin, melanin and water, as well as structural properties in skin tissue, at two imaging depths.

The study participants mainly consist of a prospective primary care population, that undergo an investigation (including SFDI assessment) at a primary care visit. Other assessment data collected during the visit (including medical history, blood pressure, blood values, ankle-brachial index) is retrieved from the participant's medical journal. An extended examination (including SFDI assessment with addition of a 3-minute post-occlusive hyperemia (PORH) test and vascular assessment using the reference system Perimed Periflux 6000) will be offered to participants based on increased risk of cardiovascular disease in the primary care population, or for separately invited subjects with increased cardiovascular risk, known diabetes or as healthy controls. Repeated yearly measurements may be performed in subjects who are interested in doing so.

A subset of participants will undergo a multi-modal investigation which includes combining data from the current study with contactless laser vibrometry data from the investigation "Cardio Alpha" (CIV ID: CIV-22-08-040426). The hypothesis is that cardiovascular disease (CVD) risk assessment may be improved through a multi-modal approach, combining data on both macro- and microcirculatory function.

Another subset of participants will undergo a diabetic feet assessment protocol, including an SFDI assessment of the soles of the feet and assessment using reference methods for macro-and microcirculation, and a foot neuropathy assessment.

A third subset of participants will undergo a skin cancer assessment protocol, including SFDI assessment of a suspected lesion on the skin.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients part of the regular healthcare patient flow at the investigational sites, or as separately invited to participate in this investigation.
* Patients with signed informed consent

Exclusion Criteria:

* Cognitive impairment
* Patients unable to understand the oral and written study information in Swedish or English
* Other severe disorder or terminal disease
* Patients unable to provide an informed consent
* Patient´s with damaged, scarred or non-intact skin within the skin area of interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study participants mainly consist of a prospective primary care population. All patients visiting the clinical sites, seeking care, or as separately invited, are offered to participate in this investigation. This includes sub-groups of patients with conditions such as diabetes mellitus, peripheral arterial disease and skin cancer. An extended investigation will be offered to participants judged to have an increased risk of cardiovascular disease in the primary care population, or for separately invited subjects with increased cardiovascular risk, or as healthy controls. Repeated yearly measurements plan to be performed in interested subjects.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Association between IMD-derived variables and markers for circulatory deficiencies measured by CE-marked reference systems | Same day as enrolment, or typically within 3-6 months from enrolment. If 1-year follow-up, then 1 year and 3-6 months from enrolment.
  Evaluate the correlation between IMD-derived parameters and outcomes related to vascular function, including ankle-brachial index, toe-brachial index and tcpO2, acquired by CE-marked reference system Perimed® Periflux 6000 or CE-marked oscillometric ABI measurement device.
Performance of a combined risk score using data from Spectrum 1 and the in parallel performed investigation "Cardio Alpha"(CIV-ID: CIV-22-08-040426) | Same day as enrolment or typically within 3-6 months following enrolment. If 1-year follow-up, then typically 1 year and 3-6 months from enrolment.
  Assess performance in prediction of cardiovascular disease risk when adding parameters from the clinical study "Cardio Alpha" to parameters from the present study. Outcomes will include known CVD or CVD risk, based on established risk factors, risk scores, clinical information and outcomes from reference devices from both investigations.

SECONDARY OUTCOMES:
Association between peak oxygen saturation measured by spatial frequency domain imaging (SFDI) on the palm and forearm and cardiovascular risk factors. | Typically 3-6 months from enrolment. If 1-year follow-up, then 1 year and 3-6 months from enrolment.
  To evaluate the association between peak oxygenation obtained from the investigational device upon release of a 3-minute post-occlusive hyperemia (PORH) test, and established CVD risk factors, including brachial blood pressure, BMI, hypertension diagnosis, diabetes mellitus diagnosis, smoking status, hsCRP and HbA1C, in a large cohort within primary care.
Correlation between oxygenation on sole of the foot and tissue ischemia level | Same day as enrolment.
  To evaluate correlation between markers of oxygenation (oxygen conc., total hemoglobin conc., oxy-and deoxy-hemoglobin conc.) on the foot sole and transcutaneous oxygen pressure (tcpO2), acquired using Perimed® Periflux 6000 reference device, in diabetic subjects.
Correlation between oxygenation on sole of the foot and neuropathy | Same day as enrolment.
  To evaluate the correlation between markers of oxygenation (oxygen conc., total hemoglobin conc., oxy-and deoxy-hemoglobin conc.) on foot sole and degree of neuropathy assessed by VibroSense® Meter II neuropathy score, in diabetic subjects.
Correlation between water concentration on sole of the foot and tissue ischemia level | Same day as enrolment.
  Regression coefficient from correlation between water concentration within measured volume on foot sole and transcutaneous oxygen pressure (tcpO2), acquired using Perimed® Periflux 6000 reference device
Correlation between water concentration on sole of the foot and neuropathy | Same day as enrolment.
  Regression coefficient from correlation between melanin and water concentration within measured volume on foot sole and degree of neuropathy assessed by VibroSense® Meter II neuropathy score.
Difference in oxygenation/ hemoglobin gradient between lesion and surrounding tissue | At follow-up, within 3 months of enrolment.
  Relative gradient in oxy- and deoxy-hemoglobin concentration, total hemoglobin concentration and/or oxygen concentration in malignant and non-malignant skin lesions compared to surrounding tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Rodgers, MD, Principal Investigator — HJN Sverige AB/Neko Health AB
Locations (3):
- Sweden (3):
  - Atrium Health Care Centre, Stockholm
  - Neko Health Centre, Regeringsgatan, Stockholm
  - Neko Health Centre, Sibyllegatan, Stockholm

IPD SHARING:
Plan to Share IPD: No